CLINICAL TRIAL: NCT06231797
Title: AI-ECG Screening for Left Ventricular Systolic Dysfunction: A Prospective, Observational, Multicenter Study
Brief Title: AI-ECG Screening for Left Ventricular Systolic Dysfunction
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: H-2306-083-1439
Record Dates: First submitted 2023-11-02; First posted 2024-01-30 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2023-10

CONDITIONS: Left Ventricular Systolic Dysfunction
MeSH Terms: conditions — Ventricular Dysfunction, Left | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: AI algorithm conducted on 12-lead ECG and transthoracic echocardiography — 12-lead ECG is performed for each patient. For 12-lead ECG, AITIALVSD (AI algorithm) analysis will be performed through a separate server.

SUMMARY:
The purpose of the current study is to verify the effectiveness of the artificial intelligence algorithm applied to the electrocardiogram as a potential screening tool for left ventricular systolic dysfunction.

DETAILED DESCRIPTION:
The current investigators have developed an artificial intelligence (AI) algorithm based on 12-lead electrocardiogram (ECG) detecting left ventricular systolic dysfunction, through 364,845 ECGs from 148,547 patients. Then, when the model was tested retrospectively on 59,805 ECGs of 24,376 patients, the model performance expressed as an area under the receiver operating characteristic curve was 0.889 (95% CI 0.887-0.891).

The investigators are planning to prospectively validate the model's effectiveness as a potential screening tool for left ventricular systolic dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Individuals or those whose legal representative agree to participate in the study, and sign the consent form
* Can complete both 12-lead electrocardiogram and transthoracic echocardiography

Exclusion Criteria:

* Individuals whose age is less than 18 year-old.
* Individuals who do not agree to participate in the study
* Patients who are unable to participate in clinical trials at the discretion of the investigator

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing 12-lead ECG and transthoracic echocardiography in routine clinical practice
Sampling Method: Non-Probability Sample
Enrollment: 1530 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-07-10 (Estimated); Study Completion 2025-07-10 (Estimated)

PRIMARY OUTCOMES:
Area under the receiver operating characteristic curve (AUROC) | Through study completion, an average of 1 year
  AI model performance detecting LVSD, expressed as an AUROC. As a diagnostic assistance for LVSD, an ROC curve expressed as sensitivity to (1-specificity) will be presented, and the accuracy of prediction will be confirmed by calculating the AUROC, which is the area below.

SECONDARY OUTCOMES:
Sensitivity | Through study completion, an average of 1 year
  AI model sensitivity detecting LVSD
Specificity | Through study completion, an average of 1 year
  AI model sensitivity detecting patients with normal left ventricular systolic function
Positive predictive value | Through study completion, an average of 1 year
  Positive predictive value in the recruited patient population
Negative predictive value | Through study completion, an average of 1 year
  Negative predictive value in the recruited patient population

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Pyo Lee, MD, PhD, Principal Investigator — Seoul National University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kwon JM, Jo YY, Lee SY, Kang S, Lim SY, Lee MS, Kim KH. Artificial Intelligence-Enhanced Smartwatch ECG for Heart Failure-Reduced Ejection Fraction Detection by Generating 12-Lead ECG. Diagnostics (Basel). 2022 Mar 8;12(3):654. doi: 10.3390/diagnostics12030654. PMID 35328207
- [Result] Kwon JM, Kim KH, Jeon KH, Kim HM, Kim MJ, Lim SM, Song PS, Park J, Choi RK, Oh BH. Development and Validation of Deep-Learning Algorithm for Electrocardiography-Based Heart Failure Identification. Korean Circ J. 2019 Jul;49(7):629-639. doi: 10.4070/kcj.2018.0446. Epub 2019 Mar 21. PMID 31074221